CLINICAL TRIAL: NCT04228315
Title: Identification of Hypnozoite Biomarkers and Relapse Patterns of Plasmodium Vivax
Brief Title: Biomarkers of P. Vivax Relapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Armed Forces Research Institute of Medical Sciences, Thailand (Other Government)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WR2643
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-12

CONDITIONS: Malaria; Vivax Malaria; Relapse; CYP2D6 Polymorphism
Keywords: primaquine; biomarker; hypnozoite; efficacy
MeSH Terms: conditions — Malaria; Malaria, Vivax; Recurrence | interventions — Primaquine

STUDY DESIGN:
Intervention Model Description: The clinical study is a two arm, randomized, open-label treatment study of Thai adults with acute infection with P. vivax. All subjects will be treated with a short acting oral antimalarial, artesunate, to eradicate P. vivax malaria from the bloodstream. Radical cure with primaquine (15 mg/ day for 14 days) to eliminate the relapsing hypnozoite of P. vivax will be given at different times, depending on this study arm. Ten healthy controls will also be enrolled for 1 day to provide baseline samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early primaquine group (Experimental): Thirty (30) P. vivax-infected adults will be enrolled in Khun Han Hospital to receive 5 days or oral artesunate (4 mg/kg) and 15 mg/day of oral primaquine for 14 days
  Interventions: Drug: Primaquine
- Delayed Primaquine group (Active Comparator): Sixty (60) P. vivax-infected adults will be enrolled in Khun Han Hospital to receive 5 days or oral artesunate (4 mg/kg) and the primaquine regimen (15 mg/day for 14 days) not given until 42 days after enrollment
  Interventions: Drug: Primaquine
- Healthy control group (No Intervention): Ten (10) age- and gender-matched controls will be enrolled for one day to obtain biological samples to be compared to the 2 intervention arms

INTERVENTIONS:
Drug: Primaquine — radical cure dosing
  Arms: Delayed Primaquine group; Early primaquine group

SUMMARY:
Plasmodium vivax malaria is difficult to manage because even after taking medicine that kills the infection in the blood, it can continue to hide quietly in the liver, later re-emerging into the blood and causing another episode of malaria illness (relapse). This clinical trial aims to enroll patient with P. vivax infections and try to detect signals in blood, urine and/or saliva coming from the silent liver stages to help identify who could benefit from treatment with primaquine. It also will explore if certain factors of patients negatively impact primaquine efficacy.

DETAILED DESCRIPTION:
Plasmodium vivax, the most widely distributed human malaria, has resisted control largely due to a relapsing hypnozoite liver stage that is clinically silent until emergence and replication in the blood weeks to months later. Curative treatment with primaquine is often not achieved due to potential toxicity in those with G6PD deficiency, poor adherence to the two-week course, and ineffective metabolism of primaquine in those with polymorphisms in cytochrome P450 isoenzyme 2D6 (CYP2D6). Identifying those who harbor hypnozoites will allow for judicious use of primaquine in returning travelers/active duty personnel as well as targeted administration to those living in endemic areas to interrupt parasite transmission in the community. The trial will be conducted in patients presenting with uncomplicated P. vivax malaria at clinical trial sites run by Armed Forces Research Institute of Medical Sciences (AFRIMS) in Southeast Asia. It is designed to capture vivax patients who still harbor the dormant liver stage hypnozoites after treatment with a short acting oral blood schizonticide, and subsequently relapse during the follow-up period while staying in in study-provided housing to reduce risk of reinfection and surveilled daily for parasites or clinical signs of relapse. Longitudinal blood and urine sampling will be done to allow for retrospective analysis to identify biomarkers of hypnozoite infection and subsequent relapse using a systems biology approach. A smaller arm will be enrolled and will receive the short-activing schizonticide with primaquine radical cure at time of admission and followed similarly for relapse. All subjects will be followed for a total of 6 months in order to assess effectiveness of primaquine radical cure for P. vivax infections.

ELIGIBILITY:
Inclusion Criteria:

For P. vivax-infected malaria subjects

1. Are a Thai male or non-pregnant/non-lactating female aged at least 18 years and are able to fluently speak and understand Thai
2. Willingness to participate in the study as evidenced by witnessed, signed informed consent from the subject (written or thumb print)
3. Have P. vivax malaria mono-infection as determined by blood smear, with a parasitemia range of 100-400,000 parasites/microliter
4. Are available to stay in a controlled setting for the first 28 days of this study to minimize exposure to mosquitoes and available for follow-up for anticipated study duration
5. Resides in Sisaket or Ubon Ratchathani Province
6. Are of normal (non-deficient or >30% activity) G6PD phenotype as defined by WHO
7. Agree to not seek outside medical care prior to contacting the Armed Forces Research Institute of Medical Sciences (AFRIMS) study team if a fever develops during study participation (approximately 180 days), unless emergency medical care is required

For healthy control group

1. Are a Thai male or non-pregnant/non-lactating female aged at least 18 years and are able to fluently speak and understand Thai
2. Willingness to participate in the study as evidenced by witnessed, signed informed consent from the subject (written or thumb print)
3. Free of malaria and other significant health problems as established by medical history, laboratory assessment and clinical examination by clinical investigator
4. Normal (non-deficient or > 30% activity) G6PD phenotype as defined by World Health Organization (WHO)
5. Resides in Sisaket or Ubon Ratchathani Province

Exclusion Criteria:

For P. vivax-infected malaria subjects

1. Have an allergic reaction to artesunate or primaquine
2. History of anti-malarial drug use within the past 28 days
3. Have symptoms of severe malaria needing urgent treatment, such as serious vomiting, unable to eat or drink, prostration, or other signs/symptoms of concern to the doctors
4. Are a pregnant or lactating female, or female of childbearing age, up to 50 years of age or otherwise individually assessed for childbearing potential, who does not agree to use an acceptable form of contraception (e.g. pills or injectable) during this study and for 1 month after study completion
5. Chronic use of medications known to cause drug interactions with primaquine or CYP450 2D6 (selective serotonin reuptake inhibitors (SSRIs) or other medications used for psychological conditions, as well as antihistamines, antihypertensives, codeine)
6. Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study

For healthy control group

1. Has history of malaria infection in the past 10 years
2. Positive for any Plasmodium species by blood smear or PCR at time of screening
3. Pregnant or lactating female
4. G6PD deficient as defined by WHO
5. Any other significant finding that in the opinion of the investigator would increase the risk of compromising the validity of being a control (eg., chronic daily chewing of betel nut (may impact saliva assays) or menstruating females (whereby urine collections may have blood and impact assay results), etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Therapeutic efficacy of a radical cure course of primaquine for uncomplicated P. vivax infection | 6 months
  In subjects presenting with uncomplicated P. vivax infection, determine frequency of P. vivax recurrence throughout the study period after being administered a 14-day course of primaquine
Build a biorepository of prospectively collected blood and urine samples in P. vivax patients prior to relapse to analyze for hypnozoite biomarkers | 6 months
  At pre-determined time points, collect biological samples to be processed and stored for proteomic, metabolomic, genomic and transcriptomic markers of latent hypnozoites, allowing for comparisons of markers in those who did and those who did not relapse

SECONDARY OUTCOMES:
Characterize the patterns of relapsing Southeast Asian P. vivax in infected subjects | 28 days
  Percentage of P. vivax relapse in subjects with uncomplicated P. vivax mono-infection in the 28 days following treatment with oral blood stage anti-malarial treatment with comparisons between those administered primaquine at enrollment and those who did not receive primaquine
Delineate relapse kinetics of P. vivax infection using molecular diagnostic methods, | 42 days
  At pre-determined time points starting at admission and prior to P. vivax relapse, compare limit of detection of recently emerged erythrocytic forms by blood smear, polymerase chain reaction (PCR) and ultra sensitive PCR
Determine percentage of P. vivax isolates resistant to antimalarial drugs used for treatment | 6 months
  Parasite growth inhibition as measured by concentration at which 50% of growth is inhibited (IC50) to antimalarial drug panel using pLDH ELISA techniques
Establish rates of P. vivax relapse versus new infection with vivax using molecular methods | 6 months
  Perform genome sequencing to determine genetic signatures of the vivax parasite, comparing initial infection with recurrences to identify relapse versus a new infection
Characterize the rate glucose 6-phosphate dehydrogenase (G6PD) deficiency of study population | 3 months
  Incidence of G6PD deficiency (<30% activity) using quantitative spectrophotometry diagnostics
Characterize hepatic cytochrome P450 (CYP450) 2D6 enzyme genotypes and predicted phenotypes in this study population | 1 day
  Genotype CYP450 2D6 alleles in this study population and resultant predicted metabolism phenotypes using Activity Score A (AS-A)
Determine primaquine pharmacokinetics in this study population | 56 days
  Measure plasma concentrations of primaquine and its major metabolites at 0,2,4,8,10 and 24 hours after initial primaquine dose and calculate the area under the curve (AUC) for each subject
Determine primaquine pharmacokinetics in this study population | 56 days
  Measure urine concentrations of primaquine and its major metabolites at 0-4 hours, 4-10 hours and 10-24 hours after initial primaquine dose and calculate the area under the curve (AUC) for each subject
Assess impact of risk factors of travel and prior malaria history on P. vivax relapse kinetics | 6 months
  Determine number of days of travel to high malaria risk areas in 30 days prior to enrollment for each subject to compare with parasite genetic relatedness of initial and recurrent vivax infections
Measure rates of gametocyte carriage | 6 months
  Determine rate and duration of sexual stage infections based on light microscopy and molecular analyses (PCR) from samples drawn at enrollment and pre-determined time points over study period
Determine if humoral immunity contributes to protection against P. vivax recurrence | 6 months
  Measure antibody levels against vivax antigens merozoite surface protein-1 (MSP-1) and circumsporozoite protein (CSP) at Day 0,28,90 and 180 and compare to rate of P. vivax recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Norman Waters, PhD, Study Director — Armed Forces Research Institute of Medical Sciences, Thailand; Michele Spring, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand; Ladaporn Bodhidatta, MD, Principal Investigator — Armed Forces Research Institute of Medical Sciences, Thailand
Locations (1):
- Khun Han Hospital, Khun Han, Thailand